CLINICAL TRIAL: NCT04356482
Title: DETERMINATION OF THE DOSE AND EFFECTIVENESS OF CONVALESCENT PLASMA IN SEVERELY AND VERY SEVERELY ILL PATIENTS BY COVID-19
Brief Title: CONVALESCENT PLASMA FOR ILL PATIENTS BY COVID-19
Acronym: COPLASCOV19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Collaborators: SECRETARIA DE SALUD DEL ESTADO DE SONORA (Unknown); CENTRO ESTATAL DE LA TRANSFUSION SANGUINEA (Unknown); HOSPITAL CENTRAL NACIONAL PEMEX NORTE (Unknown); HOSPITAL DE ZONA No. 2 IMSS (Unknown); HOSPITAL DE ZONA No.14 IMSS (Unknown); HOSPITAL GENERAL DEL ESTADO DE SONORA (Unknown)
Responsible Party: Principal Investigator, Luis Villela, MD,MSc, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TERAPLASCOV2
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; SARS-CoV 2; Convalescence; Plasma; Doses
Keywords: covid-19; convalescent plasma doses; sars-Cov 2; treatment; response
MeSH Terms: conditions — COVID-19; Convalescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Determine the convalescent plasma dose to be administered to two groups: one severely ill (not intubated) and one very severely ill (intubated).
  Second phase: safety and efficacy of the plasma dose found in the same two types of patients.
  Interventions: Biological: convalescent plasma

INTERVENTIONS:
Biological: convalescent plasma — In phase 1, different amounts of convalescent plasma will be evaluated depending on the severity of the case.
  In phase 2, both clinical, laboratory, imaging and viral presence (effectiveness) and safety will be evaluated.
  Other Names: no apply

SUMMARY:
The present study will try to respond first in an initial phase, what is the minimum effective dose necessary of convalescent plasma for getting better in severly ill (not intubated) or very severely ill (intubated) patients.

Once the dose will be determined by each type of patient group (severely ill vs. very severely ill) has been determined, phase 2 of the study will begin, where the safety and efficacy of the use of plasma will be evaluated based on clinical, imaging and laboratory criteria.

So, our hypotheses are:

1. Is there a minimum effective dose to treat seriously ill patients with convalescent plasma with COVID-19?
2. the plasma dose with the minimum effective effect will improve the clinical, laboratory and clearance conditions of the presence of the virus in the severely ill patient?

DETAILED DESCRIPTION:
Specific objectives

1. Show the efficacy and safety of fresh plasma in different doses in severe cases and in very severe cases.
2. Assess whether fresh plasma can overcome negative prognostic factors in very severe ill patients with COVID-19 infection. These factors are age, high SOFA score, and high D-dimer.
3. To evaluate the titration of antiCOVID-19 antibodies and if its quantification is related to the therapeutic response.

The responses to drug treatments that exist in our country such as hydroxychloroquine ± azithromycin, lopinavir / ritonavir and tocilizumab (anti-IL-6) are very heterogeneous, with high cost and diverse and serious adverse events in some cases. Absent randomized-controlled studies and case series or small cohort studies have not been shown to be more effective than supportive treatments in these patients. One more factor is that intubated patients cannot swallow and these medications are for oral posology; the only way to administer is through a nasogastric tube, so we cannot assure that its absorption is as expected and that the blood levels do not reach therapeutic levels.

Therefore, we propose a treatment that in the first instance is in our hands, which has already proven to be effective in infection with highly pathogenic viruses such as Ebola virus, Lassar fever and other coronavirus infections (SARS1 in 2003, MERS 2012). With regard to convalescent plasma, two studies have recently been published, a series of 5 and another of 10 cases, seriously ill and with no response to the mentioned therapies (hydroxychloroquine ± azithromycin and lopinavir / ritonavir, among others). The outcomes in this series of cases have been reported satisfactory in most with few minimal adverse events (rash).

Since the convalescent plasma dose is very ambiguous in the case-series reported, we will try to find this dose. Therefore, in this initial phase, we divided it into two severity groups:

1. . Severe ill group, convalescent plasma dose on day 0, evaluation on day +3 and if you continue with the clinic and laboratories, a second dose of plasma may be administered. Always watching the safety always (early and late transfusion reactions). Clinical evaluation (including oxygenation) as well as laboratory (days +6, +9, +12, +15, +18, +21 to find the necessary dose for response. The patients will be evaluated and if they meet the response points, the minimum effective plasma dose will be recommended for phase 2.
2. . Very severe ill group, convalescent plasma dose day 0, with evaluation on day +3, will add another dose of plasma if there is no improvement clinic or laboratory, reevaluate day +6 and if required, apply another dose of plasma if there will be not clinical or laboratory improvement. Always watching security. It is reassessed clinically (including respiratory parameters) on days +9, +12, +15, +18 and +21, to find the minimal dose necessary. This sequential treatment will help reduce the risk of water overload and also assess the presence of transfusion lung injury syndrome or TRALI. A second phase, the dose and safety of treatment will be evaluated.

In the second phase , both early and late or B will be evaluated as follows:

to. Sever ill cases: plasma will be applied according to the dose you will find in phase 1b. Security and response will be evaluated in this phase.

b. Very sever ill cases: Plasma will be applied according to the dose you will find in phase 1b and the safety and response phase will be evaluated.

It will also be open (the study will not be blinded), it will not be randomized, and it will be controlled only by the severity of the patient and their characteristics of the disease (severe vs. very severe), as well as being controlled by the amount of infusion of plasma (minimum effective dose).

SECURITY ANALYSIS

The security analysis will be between the researchers in the group and another externak group. They will analyze the first 5 patients in each group (severe and very severe), the main objective for security analysis is going to be mortality related directly to plasma infusion. Subsequently, every 20 patients in each group for phase 2 will be analyzed for safety and response.

ELIGIBILITY:
Inclusion Criteria:

All patients with COVID-19 test positive and... Severe ill patient

1. Respiratory difficulty
2. Sat O2 <93% without O2 but improves with the use of supplemental oxygen
3. CT scan image: COVID-19 compatible pneumonia
4. one or more of at least: SOFA = 0 D-dimer ≥500 Age ≥ 65 years Comorbidities such as high blood pressure, diabetes mellitus type I and II, chronic kidney failure, controlled or cured cancer, ≥ 1 degree of obesity

Very severe ill:

1. Respiratory difficulty that does not improve with supplemental oxygen, requiring intubation and connecting to ventilatory support of no more than 72hrs or 3 days.
2. CT image: COVID-19 compatible pneumonia
3. one or more of at least: SOFA ≥1 Dimer D ≥ 750 Age ≥ 65 years Comorbidities such as hypertension, diabetes mellitus type I and II, Chronic Kidney Failure, Controlled or cured cancer, ≥ 1 degree of obesity.
4. Survival over 5 days.

Other inclusion criteria:

a) Pregnant women are accepted

Exclusion Criteria:

1. patients with asymptomatic/mild disease for COVID-19
2. Children less than 16 years old
3. patients with atypical pneumonia without COVID-19 diagnostic for PCR-RT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | day -1 to day +22
  no fever, respiratory improvement and blood oxygenation (Sat02, Sat02 / Fi02), general laboratory improvement.
improvement in tomographic image | day -1 to day +12
  before convalescent plasma infusion, the CT image will be compared and subsequently the evolution of images in the CT will be evaluated every 72 hours on 3 times .
test positivity for COVID-19 | day +6 to day +12
  the patients will be evaluated on three occasions the positivity of the test (PCR-RT). If two of them are negative, it will be defined as a virus-free patient.
early and late complications associated to convalescent plasma | day 0 to day +30
  Patients will be evaluated for adverse events during the plasma infusion up to 30 days after that. Especially mild and severe allergic reactions (anaphylaxis), other issues like TRALI.

SECONDARY OUTCOMES:
days at ICU | day 0 to day +30
  days of stay at ICU will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Villela, MD, Principal Investigator — ISSSTESON
Locations (3):
- Mexico (3):
  - Hospital Del Issste Regional En Guadalajara Jalisco, Guadalajara, Jalisco
  - Secretaria de Salud Del Estado de Sonora, Hospital General Del Estado, Hermosillo, Sonora
  - Hospital Central Norte Pemex, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Result] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Result] Rajam G, Sampson J, Carlone GM, Ades EW. An augmented passive immune therapy to treat fulminant bacterial infections. Recent Pat Antiinfect Drug Discov. 2010 Jun;5(2):157-67. doi: 10.2174/157489110791233496. PMID 20370679
- [Result] Keller MA, Stiehm ER. Passive immunity in prevention and treatment of infectious diseases. Clin Microbiol Rev. 2000 Oct;13(4):602-14. doi: 10.1128/CMR.13.4.602. PMID 11023960
- [Result] Burnouf T, Seghatchian J. Ebola virus convalescent blood products: where we are now and where we may need to go. Transfus Apher Sci. 2014 Oct;51(2):120-5. doi: 10.1016/j.transci.2014.10.003. PMID 25457751
- [Result] Jahrling PB, Frame JD, Rhoderick JB, Monson MH. Endemic Lassa fever in Liberia. IV. Selection of optimally effective plasma for treatment by passive immunization. Trans R Soc Trop Med Hyg. 1985;79(3):380-4. doi: 10.1016/0035-9203(85)90388-8. PMID 3898484
- [Result] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428